CLINICAL TRIAL: NCT07043764
Title: Caring Texts for Adolescents to Reduce Suicide Risk
Brief Title: Caring Contacts Via Text Message for Suicidal Adolescents After Emergency Department Discharge
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Hoffmann, Assistant Professor of Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-6680; K23MH135206 (NIH)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Suicide Prevention
Keywords: Adolescent; Text Messaging
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Treatment as usual consists of a suicide risk assessment during the emergency department visit, determination of disposition, safety planning, provision of crisis resources, and coordination of follow-up mental health services if indicated.
- Caring Contacts (Experimental): In addition to Treatment as Usual, participants will receive Caring Contacts, consisting of brief, hopeful, supportive text messages.
  Interventions: Other: Caring Contacts Text Messages

INTERVENTIONS:
Other: Caring Contacts Text Messages — Caring Contacts are brief, hopeful, supportive text messages.
  Arms: Caring Contacts

SUMMARY:
The goal of this pilot clinical trial is to learn if Caring Contacts (brief, hopeful, supportive text messages) can be delivered to adolescents with suicidal thoughts or behaviors after discharge from the emergency department, and to understand if adolescents find it acceptable to receive Caring Contacts. Researchers will also begin to explore how suicidal thoughts and behaviors change over time among participants who receive Caring Contacts along with treatment as usual, compared to participants who only receive treatment as usual.

All participants will be invited to answer survey questions when they first enroll in the study and 1, 3, 6, and 12 months after their emergency department visit. Some participants will receive Caring Contacts (brief, hopeful, supportive text messages) after their emergency department visit. Some participants will be invited to complete an interview about their experiences receiving Caring Contacts.

ELIGIBILITY:
Inclusion Criteria:

* 12 to <18 years of age
* Present to the emergency department with suicidal thoughts or behaviors as indicated by the Ask Suicide-Screening Questions (ASQ)
* Have a cell phone that can receive text messages
* Proficient in English
* Anticipated disposition of discharge from the emergency department

Exclusion Criteria:

* In care of the Department of Children and Family Services
* Unable to participate meaningfully in assent, assessments, or the intervention, as determined by the treating clinician, including any of the following: acute or chronic cognitive impairment, acute psychosis, current severe agitation, current alcohol or drug intoxication

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) Self-Report Recent | Baseline, 1 Month, 3 Months, 6 Months, 12 Months
  The Columbia-Suicide Severity Rating Scale (C-SSRS) Self-Report Recent measures recent suicidal ideation and behavior on a scale of 0-5, with higher scores indicating greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A. Hoffmann, MD, MS, Principal Investigator — Ann & Robert H. Lurie Children's Hospital of Chicago, Northwestern University
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the NIMH Data Archive
Time Frame: Data will be made available 1 year after completion of the study
Access Criteria: Approval by NIMH Data Archive
URL: https://nda.nih.gov/